CLINICAL TRIAL: NCT01815619
Title: Single-operator Cholangioscopy-guided Biopsy of Bile Duct Strictures: Randomized Trial of Evaluation of Specimens (SOCRATES)
Brief Title: Comparison of On-Site Versus Off-Site Evaluation of Cholangioscopy-Guided Biopsies of the Bile Duct
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 409832
Record Dates: First submitted 2013-02-26; First posted 2013-03-21 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Bile Duct Stricture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- on-site evaluation of specimens by cytopathologist (Experimental): The specimen will be evaluated onsite by a cytopathologist during the procedure to render a diagnosis
  Interventions: Other: on-site specimen evaluation
- off-site specimen evaluation (Active Comparator): The specimen will be evaluated offsite by a cytopathologist during the procedure and render a diagnosis
  Interventions: Other: off-site specimen evaluation

INTERVENTIONS:
Other: on-site specimen evaluation — The specimen will be evaluated on-site by a cytopathologist during the procedure to render a diagnosis
  Arms: on-site evaluation of specimens by cytopathologist
Other: off-site specimen evaluation — The specimen will be evaluated off-site by a cytopathologist
  Arms: off-site specimen evaluation

SUMMARY:
This study will test two different methods for processing biopsy specimens taken from the bile duct. Patient;s who are asked to participate int his study have a stricture in the bile duct that needs a single operator cholangioscopy-guided biopsies during endoscopic retrograde cholangiopancreatography (ERCP) so that a diagnosis can be made. Standard of care includes performing single operator cholangioscopy-guided biopsies in the bile duct and sending the tissue to the lab for testing to make a diagnosis. Using this method the investigators can establish a diagnosis only about 50% of the time. The investigators believe that if a cytopathologist is available in the endoscopy suite during the procedure to evaluate the biopsy specimens onsite, the investigators can improve the diagnostic accuracy. The purpose of this study is to compare two methods for processing biopsies obtained from the bile duct (Onsite vs. Offsite).

DETAILED DESCRIPTION:
The diagnostic accuracy rate of single operator cholangioscopy-guided biopsy is only 50%. This translates to the need for performing repeat procedures to establish a diagnosis and therefore delays patient treatment. The biopsy specimen obtained at cholangioscopy are usually processed offsite in the pathology lab. We believe that if a pathologist can assess the tissue sample during the procedure itself (onsite) and provide feedback, the diagnostic accuracy rate will improve. This translates to better (faster) diagnosis and early treatment. Therefore, we will be comparing onsite versus offsite evaluation of bile duct biopsy specimens to determine which method yields a better diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Suspected biliary stricture

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Altered surgical anatomy
* Irreversible elevation in INR > 1.5 or low platelet count < 50,000

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-02; Primary Completion 2020-04 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of cholangioscopy-directed biopsies of bile duct strictures | up to18 months
  The primary endpoint of the study is to compare the diagnostic accuracy rates between two different methods used for processing specimens obtained from the bile duct.

SECONDARY OUTCOMES:
Specimen evaluation | up to18 months
  The secondary endpoint of the study is for specimen evaluation results deemed as malignant; benign; suspicious; atypical, or non-diagnostic.
Operating characteristics | up to18 months
  The secondary endpoint of the study is to assess the operating characteristics through review of the sensitivity, specificity, negative predictive value and positive predictive value between the on-site group and the off-site group.
Costs difference between the onsite and offsite procedures | up to 18 months
  The secondary endpoint of the study is to review and compare total costs of the onsite group in comparison to the total costs of the off-site group.
Number of biopsies to achieve diagnosis | up to 18 months
  The secondary endpoint of the study is to compare between on-site and off-site specimen for the number of biopsies to achieve diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bang JY, Navaneethan U, Hasan M, Sutton B, Hawes R, Varadarajulu S. Optimizing Outcomes of Single-Operator Cholangioscopy-Guided Biopsies Based on a Randomized Trial. Clin Gastroenterol Hepatol. 2020 Feb;18(2):441-448.e1. doi: 10.1016/j.cgh.2019.07.035. Epub 2019 Jul 24. PMID 31351135
- [Derived] Navaneethan U, Hasan MK, Kommaraju K, Zhu X, Hebert-Magee S, Hawes RH, Vargo JJ, Varadarajulu S, Parsi MA. Digital, single-operator cholangiopancreatoscopy in the diagnosis and management of pancreatobiliary disorders: a multicenter clinical experience (with video). Gastrointest Endosc. 2016 Oct;84(4):649-55. doi: 10.1016/j.gie.2016.03.789. Epub 2016 Mar 16. PMID 26995690